CLINICAL TRIAL: NCT02405000
Title: Improving Trans-oral Surgical Outcomes Through Intra-operative Image Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Joseph A. Paydarfar, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D14189
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoperative CT imaging (Experimental)
  Interventions: Other: Intraoperative CT imaging

INTERVENTIONS:
Other: Intraoperative CT imaging — Intraoperative CT scan of the upper aerodigestive tract during laryngoscopy procedure

SUMMARY:
The objective of this research is to perform a pilot study on patients undergoing laryngoscopy for diagnostic and tumor staging purposes (for pharyngeal or laryngeal cancer) in which intraoperative CT imaging will be performed both prior to (but after induction of general endotracheal anesthesia) and during placement of the laryngoscope in order to better understand anatomic changes that occur during instrumentation of the oral cavity and oropharynx. The goals of the study are:

1. Develop a suite of de-identified images and surface renderings that qualitatively show how a tumor and the upper aerodigestive tract anatomy deform during a laryngoscopic evaluation.
2. Create deformation models of the upper aerodigestive tract.

This data to be used for future retractor development as well as for virtual image guided surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) seen in the Head and Neck Tumor Clinic who will require laryngoscopy in the operating room for diagnosis and staging of known or suspected tumors of the upper aerodigestive tract.

Exclusion Criteria:

* Patients who are unable to tolerate general anesthesia.
* Patients who are felt to be a "difficult airway" for induction of general endotracheal anesthesia.
* Patients with excessive dental restorations and amalgam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Radiographic evidence of upper aerodigestive tract deformation during laryngoscopy | Collected at the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Paydarfar, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided